CLINICAL TRIAL: NCT03854981
Title: Role of Pre-operative Exercise and Nutrition Therapy on Insulin Resistance and Vascular Health in Patients Undergoing Bariatric Surgery
Brief Title: Pre-operative Exercise and Nutrition Therapy on Cardio-metabolic Health in Patients Undergoing Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Steven K. Malin, PhD, Assistant Professor, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18316
Record Dates: First submitted 2019-01-24; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Bariatric Surgery Candidate
Keywords: Insulin Resistance; Cardiovascular Risk; Inflammation; Exercise; Diet
MeSH Terms: conditions — Insulin Resistance; Inflammation; Motor Activity | interventions — Exercise; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Placebo Comparator): If subjects are assigned to this group they will not be provided materials to increase exercise participation. Subjects will however be asked to participate in the standard education sessions that are provided to all bariatric surgery patients. This standard care includes meetings with a nutritionist, psychologist, and bariatric surgeon.
  Interventions: Procedure: Standard Care
- Exercise + Standard Care (Active Comparator): Subjects will be asked to exercise 5 days/week for 30 min/day at an intensity of 65-85% of their measured HRmax. Walking will be the main type of exercise. In addition to this training program, subject's will participate in the standard education sessions that are provided to all bariatric surgery patients.
  Interventions: Behavioral: Exercise; Procedure: Standard Care

INTERVENTIONS:
Behavioral: Exercise — Subjects will be asked to exercise 5 days/week in addition to receiving standard care before bariatric surgery.
  Arms: Exercise + Standard Care
Procedure: Standard Care — Standard preoperative care of bariatric surgery

SUMMARY:
Obesity is a major health concern that has been associated with an estimated 2.8 million deaths worldwide each year. The number of individuals considered obese with a Body Mass Index (BMI) above 30 kg/m2 has grown to more than 500 million. The increased morbidity and mortality associated with obesity stems from a long list of comorbidities, including hypertension, coronary artery disease, stroke, cancer, and type 2 diabetes (T2D). Bariatric surgery is an emerging intervention that has been used frequently to induce weight loss for obese individuals and it has been shown to improve glycemic control and insulin resistance in people at risk for type 2 diabetes. Surgery may also lead to healthy improvements in inflammation, immune cells and vascular health. It is already known that exercise and weight loss from lifestyle modification can improve glycemic control, insulin resistance, inflammation, and arterial stiffness. However, no work has been done to examine a combination of bariatric surgery and pre-surgery exercise. Recent work by the team has evidence demonstrating that health status pre-surgery has an impact on post-surgery outcomes. Such findings suggest that improvements in health status from exercise before surgery may improve surgery outcomes as well as surgery-induced health outcomes. To date, no study has systematically examined the role of exercise on the prevalence of surgery complications or on post-surgery weight loss, glycemic control, and insulin resistance. Moreover, no work currently exists on exercise, with or without bariatric surgery on adipose tissue derived inflammation. Therefore, the purpose of this study is to investigate the effect of pre-surgery lifestyle intervention with exercise on bariatric surgery outcomes. To test this objective, subjects will participate in a match paired study, based on BMI. Subjects will undergo testing of blood chemistry and related measures of health before (pre-test) and after (post) intervention. Then all subjects will receive bariatric surgery. Post surgery outcomes will be assessed by examining surgery operating time, changes in blood chemistry, adipose tissue biopsies and other measures indicative of glucose and vascular health. After this surgery, subjects will return for testing about 30d later.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 18-70 years of age
* BMI >30 and <70 kg/m2
* Sedentary (Not currently participating in exercise training: >30 min. of physical activity per day, >3 days/week)
* HCT for women > 36%, Men >38%
* Non-pregnant (women).-self reported
* Smoker (if bariatric surgery patient) or non-smoker (enrolled for the dietary portion of the study)
* Has the ability/willingness to participate in the study and agree to any of the arms involved in the study.
* No prior surgical procedure for obesity with the exception of a laparoscopic adjustable gastric banding (LAGB) under the condition that the band had not been adjusted in less than or equal to 1 year

Exclusion Criteria:

* Currently participating in exercise training: >30 min. of physical activity per day, >2 days/week)
* Cigarette smoking (presently or in the past 6 months), drug or alcohol abuse
* Pregnancy or breastfeeding
* History of congestive heart failure, ischemic heart disease, severe pulmonary disease.
* History of cancer (within 5 years)
* Diagnosed as insulin-dependent diabetes.
* Change in psychotropic medication dosage in past six weeks
* AST or ALT > 3 times normal range
* Currently involved in any active weight loss treatment program (other than self-directed attempt at calorie restricting diet) or lean patients (BMI <29 kg/m2).
* Current purging behavior occurring > once a week over the past six weeks (self-induced vomiting for weight control purposes, laxative or diuretic abuse)
* Revisional bariatric procedures including a RYGB reversal to a SG or a LAGB revision to a SG or RYGB if the band has been adjusted in greater than or equal to 1 year.
* Active psychotic illness, including bipolar affective disorders.
* Evidence of current suicidality or homicidality
* Conditions associated with significant cognitive dysfunction (e.g. dementia) or medical instability that puts the participant at risk
* Contraindication to exercise (severe/uncontrolled CVD; inability to walk 2 blocks, bone or joint problems )
* Allergy to "caine" family drugs (e.g. lidocaine).
* Currently taking active weight suppression medication (e.g. phentermine,bupropion SR, topiramate).
* On medication known to cause substantial weight gain (e.g. atypical antipsychotics such as olanzapine, sodium valproate, steroid therapy). This would not include medications commonly used in this population that usually result in only mild weight loss (e.g. SSRIs).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in Insulin Resistance | Through Study Completion, up to about 8 weeks
  Mixed Meal Tolerance Test

SECONDARY OUTCOMES:
Change in Augmentation Index in % | Through Study Completion, up to about 8 weeks
  Arterial Stiffness
Changes in Blood lipids in mg/dl | Through Study Completion, up to about 8 weeks
  Cholesterol and triglycerides
Length of Stay Post Surgery in minutes | Up to 1 week
  Recovery from surgery
Operating time in minutes | Surgical Procedure
  Length of Surgery

OTHER OUTCOMES:
Changes in blood glucose in mg/dl | Through Study Completion, up to about 8 weeks
  For the Mixed Meal Tolerance Test
Changes in blood pressure in mmHg | Through Study Completion, up to about 8 weeks
  At the Mixed Meal Tolerance Test
Body weight and height will be combined to determine BMI in kg/m^2 | Through Study Completion, up to about 8 weeks
  At the Mixed Meal tolerance Test
Concentration of adiponectin in pg/mg | Surgical Procedure
  From adipose biopsy
Concentration of leptin in pg/mg | Surgical Procedure
  From adipose biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Malin, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malin SK, Kashyap SR. Differences in Weight Loss and Gut Hormones: Rouen-Y Gastric Bypass and Sleeve Gastrectomy Surgery. Curr Obes Rep. 2015 Jun;4(2):279-86. doi: 10.1007/s13679-015-0151-1. PMID 26627222
- [Background] Malin SK, Bena J, Abood B, Pothier CE, Bhatt DL, Nissen S, Brethauer SA, Schauer PR, Kirwan JP, Kashyap SR. Attenuated improvements in adiponectin and fat loss characterize type 2 diabetes non-remission status after bariatric surgery. Diabetes Obes Metab. 2014 Dec;16(12):1230-8. doi: 10.1111/dom.12376. Epub 2014 Sep 14. PMID 25132119
- [Background] Shada AL, Hallowell PT, Schirmer BD, Smith PW. Aerobic exercise is associated with improved weight loss after laparoscopic adjustable gastric banding. Obes Surg. 2013 May;23(5):608-12. doi: 10.1007/s11695-012-0826-6. PMID 23196991
- [Background] Coen PM, Tanner CJ, Helbling NL, Dubis GS, Hames KC, Xie H, Eid GM, Stefanovic-Racic M, Toledo FG, Jakicic JM, Houmard JA, Goodpaster BH. Clinical trial demonstrates exercise following bariatric surgery improves insulin sensitivity. J Clin Invest. 2015 Jan;125(1):248-57. doi: 10.1172/JCI78016. Epub 2014 Dec 1. PMID 25437877
- [Background] Khanna V, Malin SK, Bena J, Abood B, Pothier CE, Bhatt DL, Nissen S, Watanabe R, Brethauer SA, Schauer PR, Kirwan JP, Kashyap SR. Adults with long-duration type 2 diabetes have blunted glycemic and beta-cell function improvements after bariatric surgery. Obesity (Silver Spring). 2015 Mar;23(3):523-6. doi: 10.1002/oby.21021. Epub 2015 Feb 3. PMID 25651277
- [Background] Mechanick JI, Youdim A, Jones DB, Garvey WT, Hurley DL, McMahon MM, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S; American Association of Clinical Endocrinologists; Obesity Society; American Society for Metabolic & Bariatric Surgery. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery. Obesity (Silver Spring). 2013 Mar;21 Suppl 1(0 1):S1-27. doi: 10.1002/oby.20461. PMID 23529939
- [Background] Malin SK, Niemi N, Solomon TP, Haus JM, Kelly KR, Filion J, Rocco M, Kashyap SR, Barkoukis H, Kirwan JP. Exercise training with weight loss and either a high- or low-glycemic index diet reduces metabolic syndrome severity in older adults. Ann Nutr Metab. 2012;61(2):135-41. doi: 10.1159/000342084. PMID 23036993
- [Background] Malin SK, Haus JM, Solomon TP, Blaszczak A, Kashyap SR, Kirwan JP. Insulin sensitivity and metabolic flexibility following exercise training among different obese insulin-resistant phenotypes. Am J Physiol Endocrinol Metab. 2013 Nov 15;305(10):E1292-8. doi: 10.1152/ajpendo.00441.2013. Epub 2013 Sep 24. PMID 24064339
- [Background] Nakamura K, Fuster JJ, Walsh K. Adipokines: a link between obesity and cardiovascular disease. J Cardiol. 2014 Apr;63(4):250-9. doi: 10.1016/j.jjcc.2013.11.006. Epub 2013 Dec 16. PMID 24355497
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Schauer PR, Burguera B, Ikramuddin S, Cottam D, Gourash W, Hamad G, Eid GM, Mattar S, Ramanathan R, Barinas-Mitchel E, Rao RH, Kuller L, Kelley D. Effect of laparoscopic Roux-en Y gastric bypass on type 2 diabetes mellitus. Ann Surg. 2003 Oct;238(4):467-84; discussion 84-5. doi: 10.1097/01.sla.0000089851.41115.1b. PMID 14530719
- [Background] Malin SK, Finnegan S, Fealy CE, Filion J, Rocco MB, Kirwan JP. beta-Cell dysfunction is associated with metabolic syndrome severity in adults. Metab Syndr Relat Disord. 2014 Mar;12(2):79-85. doi: 10.1089/met.2013.0083. Epub 2013 Nov 27. PMID 24283920
- [Background] Liu B, Kuang L, Liu J. Bariatric surgery relieves type 2 diabetes and modulates inflammatory factors and coronary endothelium eNOS/iNOS expression in db/db mice. Can J Physiol Pharmacol. 2014 Jan;92(1):70-7. doi: 10.1139/cjpp-2013-0034. Epub 2013 Oct 21. PMID 24383875
- [Background] Yassine HN, Marchetti CM, Krishnan RK, Vrobel TR, Gonzalez F, Kirwan JP. Effects of exercise and caloric restriction on insulin resistance and cardiometabolic risk factors in older obese adults--a randomized clinical trial. J Gerontol A Biol Sci Med Sci. 2009 Jan;64(1):90-5. doi: 10.1093/gerona/gln032. Epub 2009 Jan 20. PMID 19164269